CLINICAL TRIAL: NCT01037868
Title: A Randomised Trial on the Usefulness of Supportive Text Messages in the Treatment of Depressed Patients With Co-morbid Alcohol Dependency Syndrome
Brief Title: Usefulness of Supportive Text Messages in the Treatment of Depressed Alcoholics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St Patrick's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Vincent Agyapong, Assistant Professor of Psychiatry, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDublinTC
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Depression; Alcohol Use Disorder
Keywords: depression; alcohol dependency syndrome; dual diagnosis; SMS text messages
MeSH Terms: conditions — Depression; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supportive SMS messages (Experimental): Patients in the intervention group would receive twice daily supportive SMS text messages for 3 months from the treating team which would encourage/motivate them to refrain from drinking alcohol and comply with their medication. They would also receive a fortnightly phone call from an unblinded member of the research/treating team which would only serve the purpose of confirming that they still uses the mobile phone and receive the text messages.
  Interventions: Other: Supportive SMS text messages
- No supportive SMS text message (No Intervention): Patients in the non-intervention group would also receive text messages once every fortnight thanking them for participating in the study and a monthly phone call which would only serve the purpose of confirming that they still uses the mobile phone and receive the text messages.

INTERVENTIONS:
Other: Supportive SMS text messages — Patients in the intervention group would receive twice daily supportive SMS text messages for 3 months from the treating team which would encourage/motivate them to refrain from drinking alcohol and comply with their medication. They would also receive a fortnightly phone call from an unblinded member of the research/treating team which would only serve the purpose of confirming that they still uses the mobile phone and receive the text messages.
  Arms: Supportive SMS messages

SUMMARY:
Background:

There is abundant evidence that rates of comorbidity between substance use and depression are high (1, 2) and the risk of poor outcome is higher among individuals with the dual disorder compared with those with a single disorder (3, 4, 5, 6). Previous research has shown that about 50% of persons studied with severe mental illness and past substance abuse are likely to have a recurrence of substance abuse within 1 year of discharge from treatment (7).

There is therefore a clear clinical challenge in treating patients with the dual disorder which may calls for further research and the possible introduction of new and innovative strategies including the use of mobile phone technology to provide increased support for patients with the dual diagnosis.

There are established research evidence for using Short Message Service (SMS) text messages to remind patients of scheduled medical appointments (8,9,10,12, 13), coordinate medical staff,(14) deliver medical test results,(15,16) , promote smoking cessation ( 17), improve self-monitoring among the youth with type 1 diabetes( 18), promote weight loss among obese subjects (19 ) and monitor patient side effects following treatment(20).

Relevance of the research:

To date, after an extensive review of the literature using MEDLINE, Pub Med, ERIC, Web of Science, Science Direct and PsycINFO, no studies was found on the use of SMS text messages as an intervention to address abstinence amongst alcohol dependent subjects who are co-morbid for a depressive disorder. Thus, the investigators seek to determine if text messaging is a useful and effective strategy to help maintain abstinence, improve adherence with medication and ultimately promote mental stability in depressed patients discharged from an in-patient dual diagnosis programme. The investigators hypothesize that, daily supportive/reminder SMS text messages to depressed patients discharged from an in-patient dual diagnosis programme would increase alcohol abstinence rates , improve medication adherence rates and improve the overall mental well being of patients compared with those receiving treatment as usual.

DETAILED DESCRIPTION:
There is abundant evidence that rates of comorbidity between substance use and depression are high (1, 2). The risk of poor outcome is higher among individuals with both substance use and mood disorders compared with those that have a single disorder (3, 4, 5, 6). Previous research has shown that about 50% of persons studied with severe mental illness and past substance abuse are likely to have a recurrence of substance abuse within 1 year of discharge from treatment (7). In a study to evaluate the effectiveness of the dual diagnosis treatment programme established in St Patricks' Hospital in Dublin, it was discovered that 71.8% of patients achieved complete abstinence at 3 months and 55.8% at 6 months in the depression group(8).

There is therefore a clear clinical challenge in treating patients with the dual disorder which calls for further research and the introduction of new and innovative strategies capable of improving upon abstinence rates among patients. Such strategies could include the use of mobile phone technology to provide increased support for patients with the dual diagnosis which may translate into increase abstinence rates over time.

Significantly, mobile telephones are becoming integrated into virtually all aspects of society,(9,10,1112) and may provide an opportunity to improve health related behaviours , in particular through the use of Short Message Service (SMS) (13 ). In a randomized controlled trial to evaluate a text message-based intervention designed to help individuals lose or maintain weight over 4 months, the intervention group who received personalized SMS and MMS messages sent two to five times daily, printed materials, and brief monthly phone calls from a health counsellor lost more weight than the comparison group who only received only monthly printed materials (14). In another study, sending text messages to mobile phones increased the effectiveness of a smoking cessation intervention among college students (15). Similarly, in a program conducted among youth with type 1 diabetes (16), daily text messages were helpful for disease self-management, increased self-efficacy, and treatment adherence and achieved high satisfaction among participants. Again, weekly SMS self-monitoring of bulimic symptoms with automatic SMS feedback resulted in good monitoring adherence and acceptability in women aged 16 to 44 post-discharge from inpatient treatment (17). There are also established research evidence for using SMS to remind patients of scheduled medical appointments,(18,19,20,21, 22) coordinate medical staff,(23) deliver medical test results,(24,25,26) and monitor patient side effects following treatment(27).

To date, after an extensive review of the literature using MEDLINE, Pub Med, ERIC, Web of Science, Science Direct and PsycINFO, no studies was found on the use of daily text messages delivered via mobile phone as an intervention to address abstinence amongst alcohol dependent subjects who are co-morbid for a depressive disorder. Thus, we seek to determine if text messaging is a useful and effective strategy to help maintain abstinence, improve adherence with medication and ultimately promote mental stability in depressed patients discharged from an in-patient dual diagnosis programme. We hypothesize that, daily supportive/reminder SMS text messages to depressed patients discharged from an in-patient dual diagnosis programme would increase alcohol abstinence rates , improve medication adherence rates and improve the overall mental well being of patients compared with those receiving treatment as usual. Patients receiving the text messages and phone calls would also report a favourable experience and an overall satisfaction with the system.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilling the Diagnostic and Statistical Manual fourth edition(DSM IV) criteria for alcohol dependence and are co-morbid for a unipolar depression and who complete the in-patient dual diagnosis treatment programme.
* Patients must have an Mini Mental State Examination (MMSE) score of at least 25
* All patients should have a mobile phone, be familiar with SMS text messaging technology and be willing to take part in the study.

Exclusion Criteria:

* Patients who do not consent to take part in the study.
* Patients who are blind, not able to read, do not have a mobile phone or are unable to use the mobile SMS technology.
* Patients who suffer from dipolar affective disorder.
* Patients with a history of psychosis or current diagnosis of psychotic disorder
* Poly-substances dependence or abuse but not misuse.
* Patients who would be unavailable for follow-up during the study period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cumulative abstinence duration which would be measured using the TLFB and collateral reports | measured at 3 months
Becks Depression Inventory Score | Measured at 3 Months

SECONDARY OUTCOMES:
Changes in gamma Glutamyl Transferase (Gamma GT) and Mean Corpuscular Volume (MCV) values from baseline | 3 months
Global Assessment of Function Score, Obsessive Compulsive Drinking Scale Scores, Alcohol Abstinence Self-Efficacy Scale Score | Measured at 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Declan McLoughlin, PhD, Study Chair — University of Dudlin Trinity College & St Patricks University Hospital; Conor Farren, PhD, Study Director — St Patrick's University Hospital; Vincent IO Agyapong, MSc MRCPsych, Principal Investigator — University of Dublin, Trinity College Dublin
Locations (1):
- St Patrick's University Hospital, Dublin, Ireland

REFERENCES:
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Kessler RC, Crum RM, Warner LA, Nelson CB, Schulenberg J, Anthony JC. Lifetime co-occurrence of DSM-III-R alcohol abuse and dependence with other psychiatric disorders in the National Comorbidity Survey. Arch Gen Psychiatry. 1997 Apr;54(4):313-21. doi: 10.1001/archpsyc.1997.01830160031005. PMID 9107147
- [Background] Brady KT, Sonne SC. The relationship between substance abuse and bipolar disorder. J Clin Psychiatry. 1995;56 Suppl 3:19-24. PMID 7883738
- [Background] Brown RA, Monti PM, Myers MG, Martin RA, Rivinus T, Dubreuil ME, Rohsenow DJ. Depression among cocaine abusers in treatment: relation to cocaine and alcohol use and treatment outcome. Am J Psychiatry. 1998 Feb;155(2):220-5. doi: 10.1176/ajp.155.2.220. PMID 9464201
- [Background] Feinman JA, Dunner DL. The effect of alcohol and substance abuse on the course of bipolar affective disorder. J Affect Disord. 1996 Feb 12;37(1):43-9. doi: 10.1016/0165-0327(95)00080-1. PMID 8682977
- [Background] McKay JR, Pettinati HM, Morrison R, Feeley M, Mulvaney FD, Gallop R. Relation of depression diagnoses to 2-year outcomes in cocaine-dependent patients in a randomized continuing care study. Psychol Addict Behav. 2002 Sep;16(3):225-35. PMID 12236457
- [Background] Dixon L, McNary S, Lehman AF. Remission of substance use disorder among psychiatric inpatients with mental illness. Am J Psychiatry. 1998 Feb;155(2):239-43. doi: 10.1176/ajp.155.2.239. PMID 9464204
- [Background] Farren CK, Mc Elroy S. Treatment response of bipolar and unipolar alcoholics to an inpatient dual diagnosis program. J Affect Disord. 2008 Mar;106(3):265-72. doi: 10.1016/j.jad.2007.07.006. Epub 2007 Aug 16. PMID 17707085
- [Background] Katz J. Machines that become us: the social context of personal communication technology. New Brunswick New Jersey: Transaction Publishers, 2003.
- [Background] Ling R. The mobile connection: the cell phone's impact on society. San Francisco: Morgan Kaufmann Publishers, 2004.
- [Background] Patrick K, Raab F, Adams MA, Dillon L, Zabinski M, Rock CL, Griswold WG, Norman GJ. A text message-based intervention for weight loss: randomized controlled trial. J Med Internet Res. 2009 Jan 13;11(1):e1. doi: 10.2196/jmir.1100. PMID 19141433
- [Background] Obermayer JL, Riley WT, Asif O, Jean-Mary J. College smoking-cessation using cell phone text messaging. J Am Coll Health. 2004 Sep-Oct;53(2):71-8. doi: 10.3200/JACH.53.2.71-78. PMID 15495883
- [Background] Franklin VL, Waller A, Pagliari C, Greene SA. A randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes. Diabet Med. 2006 Dec;23(12):1332-8. doi: 10.1111/j.1464-5491.2006.01989.x. PMID 17116184
- [Background] Bauer S, Percevic R, Okon E, Meermann R, Kordy H. Use of text messaging in the aftercare of patients with bulimia nervosa. Eur Eat Disord Rev. 2003;11:279-290
- [Background] Bos A, Hoogstraten J, Prahl-Andersen B. Failed appointments in an orthodontic clinic. Am J Orthod Dentofacial Orthop. 2005 Mar;127(3):355-7. doi: 10.1016/j.ajodo.2004.11.014. PMID 15775951
- [Background] Downer SR, Meara JG, Da Costa AC. Use of SMS text messaging to improve outpatient attendance. Med J Aust. 2005 Oct 3;183(7):366-8. doi: 10.5694/j.1326-5377.2005.tb07085.x. PMID 16201955
- [Background] Milne RG, Horne M, Torsney B. SMS reminders in the UK national health service: an evaluation of its impact on "no-shows" at hospital out-patient clinics. Health Care Manage Rev. 2006 Apr-Jun;31(2):130-6. doi: 10.1097/00004010-200604000-00006. PMID 16648692
- [Background] Vilella A, Bayas JM, Diaz MT, Guinovart C, Diez C, Simo D, Munoz A, Cerezo J. The role of mobile phones in improving vaccination rates in travelers. Prev Med. 2004 Apr;38(4):503-9. doi: 10.1016/j.ypmed.2003.12.005. PMID 15020186
- [Background] Cohen CE, Coyne KM, Mandalia S, Waters AM, Sullivan AK. Time to use text reminders in genitourinary medicine clinics. Int J STD AIDS. 2008 Jan;19(1):12-3. doi: 10.1258/ijsa.2007.007149. PMID 18275639
- [Background] Sherry E, Colloridi B, Warnke PH. Short message service (SMS): a useful communication tool for surgeons. ANZ J Surg. 2002 May;72(5):369. doi: 10.1046/j.1445-2197.2002.02411.x. No abstract available. PMID 14696592
- [Background] Pal B. The doctor will text you now; is there a role for the mobile telephone in health care? BMJ 2003;326:607.
- [Background] Tomnay JE, Pitts MK, Fairley CK. New technology and partner notification--why aren't we using them? Int J STD AIDS. 2005 Jan;16(1):19-22. doi: 10.1258/0956462052932700. PMID 15705267
- [Background] Menon-Johansson AS, McNaught F, Mandalia S, Sullivan AK. Texting decreases the time to treatment for genital Chlamydia trachomatis infection. Sex Transm Infect. 2006 Feb;82(1):49-51. doi: 10.1136/sti.2004.014381. PMID 16461603
- [Background] Weaver A, Young AM, Rowntree J, Townsend N, Pearson S, Smith J, Gibson O, Cobern W, Larsen M, Tarassenko L. Application of mobile phone technology for managing chemotherapy-associated side-effects. Ann Oncol. 2007 Nov;18(11):1887-92. doi: 10.1093/annonc/mdm354. Epub 2007 Oct 5. PMID 17921245
- [Background] Sobell MB, Sobell LC, Leo GI. Does enhanced social support improve outcomes for problem drinkers in guided self-change treatment? J Behav Ther Exp Psychiatry. 2000 Mar;31(1):41-54. doi: 10.1016/s0005-7916(00)00007-0. PMID 10983746
- [Background] Cocosila M, Archer N, Haynes RB, Yuan Y. Can wireless text messaging improve adherence to preventive activities? Results of a randomised controlled trial. Int J Med Inform. 2009 Apr;78(4):230-8. doi: 10.1016/j.ijmedinf.2008.07.011. Epub 2008 Sep 7. PMID 18778967
- [Background] R.B. Haynes, D. Sackett, G. Guyatt, P. Tugwell, Clinical Epidemiology: How to do Clinical Practice Research, Lippincott, Williams, Wilkins, Philadelphia, PA, 2005